CLINICAL TRIAL: NCT00434109
Title: Phase II Study of Sunitinib Malate Following Hepatic Artery Embolization for Metastatic Gastrointestinal Neuroendocrine Tumors
Brief Title: Phase II Study of Sunitinib Malate Following Hepatic Artery Embolization
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-14888; GA6181079 (Other: Pfizer)
Record Dates: First submitted 2007-02-09; First posted 2007-02-12 (Estimated); Results first posted 2012-09-07 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2012-07

CONDITIONS: Neuroendocrine Tumor; Islet Cell Tumor
Keywords: Carcinoid; Pancreatic; Metastatic; Neuroendocrine; Tumors; Hepatic; Artery; Embolization; Angiogenesis; Sunitinib; Malate; Sutent; Tyrosine; Kinase; Inhibitor
MeSH Terms: conditions — Neuroendocrine Tumors; Adenoma, Islet Cell; Carcinoid Tumor; Neoplasm Metastasis; Neoplasms | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sunitinib Malate and Hepatic Artery Embolizations (Experimental): Sunitinib Malate and Selective Hepatic Artery Embolizations: Sunitinib malate (Sutent) at a dose of 37.5mg. 1-3 selective hepatic artery embolizations.
  Interventions: Drug: Sunitinib malate; Procedure: Hepatic Artery Embolizations

INTERVENTIONS:
Drug: Sunitinib malate — Sunitinib malate (Sutent) at a dose of 37.5mg will be administered orally once daily on days 1-28 in a 42-day cycle. Treatment with Sutent will begin no sooner than seven days after the first hepatic artery embolization. Subsequent embolizations (if necessary) will be scheduled during scheduled Sutent treatment breaks. No fewer than seven days shall separate treatment with Sutent and scheduling of hepatic artery embolizations.
  Other Names: Sutent
Procedure: Hepatic Artery Embolizations — 1-3 selective hepatic artery embolizations will be performed at approximately 5-week intervals, based on the extent of hepatic involvement with tumor.

SUMMARY:
The purpose of this study is to decide if a medicine that slows growth of new blood vessels can be give after the embolization procedure to prevent or delay new growth of blood vessels to tumors.

DETAILED DESCRIPTION:
This is a single-center, open-label, non-randomized, prospective phase II trial. Sutent treatment will be continued until disease progression, or excessive toxicity (as determined by treating physician or primary investigator), or until a maximum of eight cycles, whichever duration is shorter.

ELIGIBILITY:
Inclusion Criteria:

* Well-differentiated metastatic carcinoid tumors and pancreatic endocrine tumors with measurable liver metastases.
* Resolution of all acute toxic effects of prior chemotherapy or radiotherapy or surgical procedures to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 3.0 grade less than or equal to 1.
* Adequate organ function as defined by the following criteria:

  1. Serum aspartate transaminase (AST; serum glutamic oxaloacetic transaminase [SGOT]) and serum alanine transaminase (ALT; serum glutamic pyruvic transaminase [SGPT]) less than or equal to 2.5 x local laboratory upper limit of normal (ULN), or AST and ALT less than or equal to 5 x ULN if liver function abnormalities are due to underlying malignancy
  2. Total serum bilirubin less than or equal to 1.5 x ULN
  3. Absolute neutrophil count (ANC) greater than or equal to 1500/microL
  4. Platelets greater than or equal to 100,000/microL
  5. Hemoglobin greater than or equal to 9.0 g/dL
  6. Serum calcium less than or equal to 12.0 mg/dL
  7. Serum creatinine less than or equal to 1.5 x ULN
  8. Prothrombin and activated partial thromboplastin time (PT and aPTT) less than or equal to 1.5 x ULN
* Eastern Cooperative Oncology Group (ECOG) Performance Status less than or equal to 2
* Informed Consent: Patients must be aware of the nature of his/her disease process and must willingly give consent after being informed of the experimental nature of therapy, alternatives, potential benefits, side-effects, risks and discomforts.

Exclusion Criteria:

* Major surgery or radiation therapy within 4 weeks of starting the study treatment.
* Prior hepatic artery embolization or chemoembolization.
* Prior treatment with a tyrosine kinase inhibitor or a vascular endothelial growth factor (VEGF) inhibitor.
* NCI CTCAE grade 3 hemorrhage within 4 weeks of starting the study treatment.
* History of or known brain metastases, spinal cord compression, or carcinomatous meningitis, or evidence of symptomatic brain or leptomeningeal disease on screening computed tomography (CT) or magnetic Resonance imaging (MRI) scan.
* Any of the following within the 6 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism.
* Ongoing cardiac dysrhythmias of NCI CTCAE grade greater than or equal to 2.
* Prolonged corrected QT (QTc) interval on baseline electrocardiogram (EKG).
* Hypertension that cannot be controlled by medications (>150/100 mm Hg despite optimal medical therapy).
* Pre-existing thyroid abnormality with thyroid function that cannot be maintained in the normal range with medication.
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness or other active infection
* Concurrent treatment on another clinical trial. Supportive care trials or non-treatment trials, e.g. Quality of Life (QOL), are allowed.
* Concomitant use of ketoconazole and other agents known to induce CYP3A4.
* Concomitant use of theophylline and phenobarbital and/or other agents metabolized by the cytochrome P450 system.
* Ongoing treatment with therapeutic doses of Coumadin (low dose Coumadin up to 2 mg by mouth (po) daily for thrombo prophylaxis is allowed).
* Pregnancy or breastfeeding. Female participants must be surgically sterile or be postmenopausal, or must agree to use effective contraception during the period of therapy. Female participants with reproductive potential must have a negative pregnancy test (serum or urine) prior to enrollment. Male participants must be surgically sterile or must agree to use effective contraception during the period of therapy.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2006-11; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Strosberg, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials Website — http://www.moffitt.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients seen at Moffitt Cancer Center with hepatic metastases from gastrointestinal neuroendocrine tumors were screened for eligibility to be enrolled in the study.
Period: Overall Study
Arm/Group | Sunitinib Malate and Hepatic Artery Embolizations
Started | 39
Completed | 21 (Patients completing the maximum eight cycles of sunitinib.)
Not Completed | 18
Not completed — Physician Decision | 9
Not completed — Adverse Event | 5
Not completed — Protocol Violation | 1
Not completed — had embolism, did not receive sunitinib | 3

BASELINE CHARACTERISTICS:
Arm/Group | Sunitinib Malate and Hepatic Artery Embolizations
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 10
Age, Customized [Median (Full Range); unit: years] | 61 [40 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Progression Free Survival (PFS) at 12 Months
Description: Kaplan-Meier analysis of PFS. Progression-free survival rate at 12 months after first embolization. PFS was defined as time from start of treatment until disease progression or death as a result of any cause. Response and progression endpoints refer specifically to hepatic metastases. Extrahepatic metastases were included for assessment of response and progression by RECIST version 1.0. Progressive Disease (PD): At least a 20% increase in the SLD of target lesions, taking as reference the smallest SLD recorded since the treatment started.
Time Frame: 12 months
Population: All participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sunitinib Malate and Hepatic Artery Embolizations
Number analyzed (Participants) | 39
percentage of participants | 66 [51 to 81]

2. Secondary Outcome: Percentage of Participants With Overall Survival (OS) at One Year
Description: Overall survival at 12 months. OS was defined as time from start of treatment until death as a result of any cause, with patients censored at the date of last follow-up if still alive.
Time Frame: 12 months
Population: All participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sunitinib Malate and Hepatic Artery Embolizations
Number analyzed (Participants) | 39
percentage of participants | 95 [88 to 100]

3. Secondary Outcome: Number of Participants With Partial Radiographic Response
Description: Objective radiographic response rate. Response and progression endpoints refer specifically to hepatic metastases. Extrahepatic metastases were included for assessment of response and progression by RECIST version 1.0. Partial Response (PR): At least a 30% decrease in the sum of longest diameter (SLD) of target lesions, taking as reference the baseline SLD.
Time Frame: 12 months
Population: All Participants
Measure: Number; unit: participants
Arm/Group | Sunitinib Malate and Hepatic Artery Embolizations
Number analyzed (Participants) | 39
participants | 28

4. Secondary Outcome: Number of Participants With Biochemical Response
Description: Biochemical response rate (>50% reduction in tumor marker). Response and progression endpoints refer specifically to hepatic metastases.
Time Frame: 12 months
Population: All Participants
Measure: Number; unit: participants
Arm/Group | Sunitinib Malate and Hepatic Artery Embolizations
Number analyzed (Participants) | 39
participants | 19

5. Secondary Outcome: Number of Participants Requiring Dose Reduction
Description: Treatment related toxicity. Participants requiring dose reductions of sunitinib to 25 mg due to side effects.
Time Frame: 12 months
Population: All participants
Measure: Number; unit: participants
Arm/Group | Sunitinib Malate and Hepatic Artery Embolizations
Number analyzed (Participants) | 39
participants | 16

6. Secondary Outcome: Percentage of Participants With Overall Survival (OS) at 4 Years
Description: Participant overall survival at 48 months. OS was defined as time from start of treatment until death as a result of any cause, with patients censored at the date of last follow-up if still alive.
Time Frame: 48 months
Population: All Participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sunitinib Malate and Hepatic Artery Embolizations
Number analyzed (Participants) | 39
percentage of participants | 59 [38 to 80]

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Sunitinib Malate and Hepatic Artery Embolizations
Serious Adverse Events (participants affected / at risk) | 3/39
Other Adverse Events (participants affected / at risk) | 38/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sunitinib Malate and Hepatic Artery Embolizations (N=39)
Hemorrhage, GI - Recturm - possibly related (Gastrointestinal disorders) | 1 (1)
Nausea and Vomiting - unrelated (Gastrointestinal disorders) | 1 (2)
Dysphagia - unrelated (Gastrointestinal disorders) | 1 (1)
Anorexia - unrelated (Gastrointestinal disorders) | 1 (1)
Obstruction, GI - Gallbladder - unrelated (Gastrointestinal disorders) | 1 (1)
Obstruction, GI - Small bowel - unrelated (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib Malate and Hepatic Artery Embolizations (N=39)
Hemoglobin (Blood and lymphatic system disorders) | 22
Neutrophils/granulocytes (Blood and lymphatic system disorders) | 19
Platelets (Blood and lymphatic system disorders) | 14
Abdominal pain (Gastrointestinal disorders) | 18
Anorexia (Gastrointestinal disorders) | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Back pain (General disorders) | 3
Constipation (Gastrointestinal disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dehydration (Gastrointestinal disorders) | 3
Dermatological (Skin and subcutaneous tissue disorders) | 2
Diarrhea (Gastrointestinal disorders) | 8
Dry skin (Skin and subcutaneous tissue disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Edema (Blood and lymphatic system disorders) | 11
Epistaxis (General disorders) | 2
Fatigue (General disorders) | 24
Fever (General disorders) | 12
Hair loss (Skin and subcutaneous tissue disorders) | 5
Headache (General disorders) | 7
Hemorrhoids (Gastrointestinal disorders) | 2
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 4
Hypertension (Cardiac disorders) | 9
Mood alterations (General disorders) | 2
Mucositis/stomatitis (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 14
Neuropathy (Nervous system disorders) | 3
Potassium (Metabolism and nutrition disorders) | 4
Palmar-plantar erythrodysesthesia (Skin and subcutaneous tissue disorders) | 19
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 2
Rhinitis (General disorders) | 3
Taste alterations (Gastrointestinal disorders) | 14
Weitht loss (Metabolism and nutrition disorders) | 2
Vomiting (Gastrointestinal disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes